CLINICAL TRIAL: NCT02778334
Title: Links Between Depression, Anxiety, Coping and Quality of Life After a Stroke: Depressive and Anxiety Symptoms and Individual Coping Strategies of the Acute Phase in the Fourth Month as a Factor Influencing Mental Health and Quality of Life
Brief Title: Links Between Depression, Anxiety, Coping and Quality of Life After a Stroke
Acronym: COPING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other); Laboratoire Psychopathologie et Processus de Santé (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: COPING
Record Dates: First submitted 2016-05-04; First posted 2016-05-19 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Stroke
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients who return home (No Intervention)
- patients who continued hospitalization in rehabilitation (Experimental)
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — Patients who accept will be seen in maintenance during hospitalization in Neuro-Vascular Unit (UNV) (T0 = 4 to 7 days post-stroke)
  At the time of the release of the UNV two groups:
  1. patients who return home and
  2. patients who continued hospitalization in rehabilitation. Depression, anxiety, quality of life and coping strategies will be assessed by self-administered questionnaires. A first phase of ambulatory (ESM / EMA) will also take place following the (UNV) output: 5 times a day for 7 days patients will respond to questions evaluating depression, anxiety and coping strategies. Patients will answer these questions via a smartphone app (issues ESM).
  Another ambulatory phase on the same model as that performed at T1 (5 times daily for 7 days) accompanied by a self-assessment of depression, anxiety, coping strategies and quality of life will made 2 months post-stroke (T2).
  The last time the study will take place 4 months after stroke onset (T3).
  Arms: patients who continued hospitalization in rehabilitation

SUMMARY:
Introduction and literature review With 130 000 cases per year in France in 2010, stroke is one of the most common neurological diseases, often leaving many disabling sequelae physical and cognitive levels (currently live 500 000 disabled following a stroke) and leading and a loss of significant autonomy in these patients. However, many stroke survivors soon find a range comparable to their previous state. Investigators can then ask ourselves about the impact of this life event in these people who apparently do not show visible effects: what about the psychological repercussions of stroke in these patients healthy; what is changed in their daily lives, particularly in their mental functioning after this brutal confrontation with their own mortality?

Objectives Our project aims to better understand the psychological repercussions of stroke in patients who quickly find a health and autonomy comparable to their previous state. The objective will be to investigate the relationship between depressive symptoms and anxiety, coping strategies and quality of life from the acute phase and during the first months after the onset of stroke. This period is particularly demanding for these patients must therefore adapt and readjust continuously: shock stroke, hospitalization in several services (intensive care, neurology, rehabilitation), back home, "new" life with the changes related stroke, resumption of a professional activity, etc ...

Our methodology will combine tools conventionally used (standardized interview, validated questionnaires) to newer, ecological and true methods (Experience Sampling Method applied by the use of a smarphone application) to assess different variables studied.

This initially be determined whether the various symptoms of the depression on the one hand and anxiety on the other hand, depending on their mode of expression (vs. outsourced internalized; ie emotional, cognitive, somatic), observed from the acute phase of stroke, are related and predict the quality of life, depression and anxiety in the longer term (four months after the stroke).

Furthermore, our study will observe if the individual coping strategies (coping) daily and evolution influence the psychological status and quality of life during the months following the stroke.

DETAILED DESCRIPTION:
Introduction and literature review With 130 000 cases per year in France in 2010, stroke is one of the most common neurological diseases, often leaving many disabling sequelae physical and cognitive levels (currently live 500 000 disabled following a stroke) and leading and a loss of significant autonomy in these patients. However, many stroke survivors soon find a range comparable to their previous state. Investigators can then ask ourselves about the impact of this life event in these people who apparently do not show visible effects: what about the psychological repercussions of stroke in these patients healthy; what is changed in their daily lives, particularly in their mental functioning after this brutal confrontation with their own mortality? Research on psychology and psychiatric disorders post-stroke indicate a frequency of occurrence of depression in 30-40% of patients, while the occurrence of anxiety disorders in 20% to 30% of patients. Depression and anxiety after stroke is influenced by the presence of sequels, but in a preliminary study (see Psycho-stroke current study) with patients with no impairment of their independence three months after stroke Investigators observed the presence of depressive and anxious symptoms.

The psychological health influences the patient's quality of life overall. Recent results have thus demonstrated that post-stroke depression increased the risk of short- and long-term mortality. It therefore seems essential to identify risk factors and influence of depression and anxiety after stroke, particularly in patients rapidly and almost completely recovering from the aftermath of their accident, to prevent the emergence and to support them.

In the scientific literature, individual coping strategies or coping strategies, and their development are identified as a factor of influence of post-stroke psychological health. Thus, an active coping centered on the problem would be associated with better mental health status, while a passive coping centered on managing emotions would instead be a poor prognostic factor. However, the clinical understanding of the everyday process of adaptation among survivors of stroke is limited by the assessment methods conventionally used in the research, which questioned the memory "in general" of the subject.

Modern techniques and increasingly used, as Experiences Sampling Method (ESM) or the Ecological Momentary Assessment (EMA) allow the assessment of individual functioning in more ecologically being carried out in the natural environment of the subject and greatly limit through retrospective recall. The application of these methods to a population of stroke survivors has already been validated and one study also shows that the active behaviors (work, sport) would be a post-stroke depression risk factor, whereas the presence of a social environment (among friends, relatives) would be a protective factor. However, this study is only interested in certain types of behavior, comparable to some coping strategies (active coping, social support research) but not representative of a whole, while other studies specifically interested in the evaluation of coping with this method but not with stroke patients. It seems interesting to use a similar methodology to observe in vivo finer and more accurate adaptation strategies in stroke survivors, and thus have an ecological representation of their coping.

The other factor of influence that Investigators chose to investigate in our study relates to the symptomatic forms of depression and anxiety. It is important first to note that the somatic and cognitive consequences of stroke are close to some depression and anxiety manifestations. This symptomatic overlap makes it difficult locating and diagnosing these disorders. Determine their specific seems necessary, and would involve the identification of symptoms of these psychopathological that would significantly associated with depression and anxiety lasting and intense.

Studies of post-stroke depression reveal that symptoms related to mood, thoughts and depressive emotions are more durable and predict diagnosis and depression intensity in the longer term, then somatic symptoms (fatigue) during the acute phase of stroke showed no significant association with long-term mental health.

Investigators found no published studies indicating the results on this subject regarding post-stroke anxiety. However, in the Psycho-stroke current study, initial results show that the psychic symptoms of anxiety three months after the stroke predicted anxiety in six months. Investigators would like to deepen these results by focusing on these shorter-term variables, that is to say from the first days after the occurrence of the accident, and study their links with the mental health status and quality life during the first months following the stroke.

Again, the use of modern evaluation methods (ESM / EMA) will capture the emotional and psychological phenomena almost instantaneously, and thus promote the clinical understanding of mental disorders after stroke. This approach, already applied in the context of post-stroke depression, however, was not used in the study of anxiety in this population, although research with d other populations are interested in anxiety as assessed.

Objectives:

Our project aims to better understand the psychological repercussions of stroke in patients who quickly find a health and autonomy comparable to their previous state. The objective will be to investigate the relationship between depressive symptoms and anxiety, coping strategies and quality of life from the acute phase and during the first months after the onset of stroke. This period is particularly demanding for these patients must therefore adapt and readjust continuously: shock stroke, hospitalization in several services (intensive care, neurology, rehabilitation), back home, "new" life with the changes related stroke, resumption of a professional activity, etc ...

Our methodology will combine tools conventionally used (standardized interview, validated questionnaires) to newer, ecological and true methods (Experience Sampling Method applied by the use of a smarphone application) to assess different variables studied.

This initially be determined whether the various symptoms of the depression on the one hand and anxiety on the other hand, depending on their mode of expression (vs. outsourced internalized; ie emotional, cognitive, somatic), observed from the acute phase of stroke, are related and predict the quality of life, depression and anxiety in the longer term (four months after the stroke).

Furthermore, our study will observe if the individual coping strategies (coping) daily and evolution influence the psychological status and quality of life during the months following the stroke.

Methodology

Population

N waited 75 patients. Recruitment Location: Neuro-Vascular Unit at St. Joseph Hospital.

Study duration: 18 to 24 months depending on the pace of inclusion.

Procedure

After submission and approval of the project by the Patient Protection Committee will be proposed to patients fulfilling the inclusion criteria to participate in the study after being informed of its progress and its objectives (note (cf. . Annexes) and meeting with the psychologist). Camille Vansimaeys, psychologist and principal investigator of this study will also be the only one to see patients and to conduct interviews as part of this research. Patients who accept will be seen in maintenance during hospitalization in Neuro-Vascular Unit (T0 = 4 to 7 days post-stroke) to assess depression and anxiety (hetero-evaluation). Socio-demographic and medical data will be collected in files and anonymous.

At the time of the release of the UNV (T1 = 12 day average hospitalization), patients will be divided into two groups: 1) patients who return home and 2) patients who continued hospitalization in rehabilitation. Depression, anxiety, quality of life and coping strategies will be assessed by self-administered questionnaires. A first phase of ambulatory (ESM / EMA) will also take place following the UNV output: 5 times a day for 7 days patients will respond to questions evaluating depression, anxiety and coping strategies. Patients will answer these questions via a smartphone app (issues ESM). The application will be directly installed on personal smartphones patients who have them. For patients who do not own a smartphone configured only to be used for the application will be lent their time to the study by the University Paris Descartes. Patients who will be entrusted these smartphones will sign an additional form framing the terms of the loan. An explanation of the operation of the application and smartphones will be made at the time of the first interview in hospital, a training phase is then performed during hospitalization.

During phase measurements by smartphones, patients will be contacted three days after the first evaluation, to address and resolve any difficulties of use, and to remind people with a smartphone lent loading.

Another ambulatory phase on the same model as that performed at T1 (5 times daily for 7 days) accompanied by a self-assessment of depression, anxiety, coping strategies and quality of life will made 2 months post-stroke (T2).

The last time the study will take place 4 months after stroke onset (T3). Patients will be reviewed in interview to assess depression and anxiety (hetero and self assessments) as well as coping strategies and quality of life (self-questionnaires). Ambulatory measurement phase (for 1 week, 5 times a day) also accompanied this evaluation. It will be made before the interview to half our population, and then the other half to control a possible parasitic effect.

ethical implications The intervention of this research with vulnerable patients by the occurrence of a stroke, and therefore may have a certain psychic and emotional vulnerability in a particularly challenging time for them, implies that Investigators are attentive to many ethical considerations.

First, it is important to emphasize that proper monitoring will be offered to patients whose psychic suffering is manifest in the different assessments. Investigators will verify if they have followed up to these difficulties, and if so Investigators redirect to health professionals so that they can be supported.

Similarly, patients who simply express a follow-up request will be directed to an appropriate care.

It will also be checked that each patient and willing to participate in this research has understood the objectives and conduct.

It will also be specified clearly that their participation, their refusal to participate or withdrawal during the study in no case affect the management or the relationship with the medical and nursing teams.

Tools

All tools used were validated their French version.

• Straight-evaluation The hetero-evaluative tools involve the identification of semiotic elements in a semi-structured clinical interview conducted by an experienced evaluator and trained in the award of these tools (in this case the clinical psychologist in charge of the study). They are not filled by patients, it is the investigator (psychologist) who asks questions based on these questionnaires, but that can be formulated differently in different patients.

MINI (Mini International Neuropsychiatric Inventory) (Sheehan et al., 1998; Lecrubier et al., 1998). This is a must-semi-structured interview guide in psychological research, the use of which is part of the professional practice of psychologist. This inventory is to gather information and semiotic elements to assist in the diagnosis of certain psychiatric disorders according to DSM-IV. Modules A (major depressive disorder), B (dysthymia), I (post-traumatic stress disorder), O (GAD) and L (psychotic disorders) MINI will be used to assess the presence or absence of disorders mood (major depression, dysthymia), anxiety disorders (generalized anxiety or post-traumatic stress, assess relevant in our study by the traumatogenic dimension of Stroke) and identify subjects which present a psychotic disorder to not to include in the study, mainly because of their altered perception of reality. In addition, the module for psychotic disorders is introduced to the patient by telling him that now the invastigator will ask him questions about some unusual or bizarre experiments that can occur in some people. "Thereby depersonalize maintenance reassurance on the fact that these issues are part of a standard valuation method and they are not raised in order to argue a diagnostic hypothesis concerning him .

MADRS (10 items) (Montgomery and Asberg Depression Rating Scale) (Montgomery and Asberg, 1979; Lempérière, 1984) will be used to assess the intensity of depressive symptoms. This scale is the reference scale in this area, it includes ten items that assess different aspects of depressive symptomatology.

HAM-A (14 items) (Hamilton Anxiety Rating Scale) (Hamilton, 1959 Pichot, 1959) is a scale for measuring state anxiety. This scale have an intensity score of general anxiety, consisting of two sub-scores for somatic anxiety one hand, and on the other psychic anxiety.

• Self evaluation These tools are questionnaires that are completed by the person who self-evaluated.

BDI-II (21 items) (Beck Depression Inventory 2nd ed) assesses the severity of depressive symptoms. Twenty-one groups of statements on the different symptoms of depression are available, the patient selects the one that best matches how he feels. The advantage of choosing this tool is that it assesses different aspects of depression both in terms of physical symptoms that cognitive and emotional.

HADS (14 items) (Hospital Anxiety Depression Scale). This scale assesses the severity of depressive and anxious symptomatology. This is the most used tool in all somatic diseases and neurological particular. This survey presents the advantage of being very short, while assessing symptoms both somatic and psychological symptomatology of these.

Brief-COPE (28 items):

This questionnaire assesses 14 separate dimensions of coping (two items per dimensions): active coping, planning, instrumental support, emotional support, expression of feelings, positive reinterpretation, acceptance, denial, blame, humor, religion, entertainment, substance use and disengagement behavioral.

WHOQOL BREF is a scale assessing the quality of life using 26 items, including two related to the overall quality of life. This questionnaire allows us to understand dimensionally the subjective perception of the person's life, in the different fields that can compose. Physical health: including aspects such as pain, fatigue or working abilities; mental health: composed among others by the positive and negative emotions and self-esteem; social relations: including personal, private life or the available social support; and finally the living environment with elements such as financial resources, access to information resources, recreation, etc ...

• Ambulatory Measures: ESM / EMA These measures will be carried out via a smartphone app. The selected items are from previous studies that measured these variables, or built specifically for the study on the basis of validated tools.

Symptoms of depression and anxiety: the symptoms of depression and anxiety present in the DSM-IV-TR and show a variability in a day will be assessed dimensionally on a Likert scale 7 points. Eg for depression: sad mood, anhedonia, fatigue, difficulty concentrating, negative / pessimistic thoughts.

Life events: questions will focus on the occurrence in the last three hours of events that have a positive impact on one hand, and negative on the other. Participants should indicate the specific areas of life for these events.

strategies to adapt to stressful events: coping strategies will be evaluated by adapting the questions brief-COPE. Participants will indicate how they reacted to the negative event previously identified by selecting from a list of statements those that match their response, for example: "I turned (e) to work or other activities to take my mind. "

Evaluation methods used at different times of the study:

Preservation and analysis of data:

A basic anonymous data will be created. Only the investigator will have access to the concordance table to link the questionnaires completed by patients with data in the database is created.

The statistical study will be conducted by the investigator himself locally in the hospital Saint Joseph group. There will be no exchange of data. Different statistical tests will be used to analyze the data: analyzes of variances, correlations, regressions. Investigators will try and update significant associations between depressive and anxious symptoms, coping and quality of life during the first months after stroke, controlling the influence variables effect (neurological status, level autonomy, hospital stay and time of return home, etc ...). Investigators will compare the evolution of different dimensions between the two subgroups of patients (back home or inpatient rehabilitation T1 service).

Medical information on stroke and data on the effects (cognitive and motor functions affected, severity of sequelae, areas in which autonomy would eventually be reduced, type and location of stroke, etc ...) will be account when analyzing the results to investigate the possible existence of links between and anxiety and depression levels.

The data stored on smartphones will be transferred directly to the smartphone to the computer that will store the data; is hosted on a secure server certified. In this case, the server will either already obtained the necessary authorizations CNIL; or an application will be made.

Expected results

The general clinical significance of this project is to determine the elements for identifying, at the time of initial hospitalization following a stroke, patients at risk of adversely psychological evolution as physical and medical condition allows them to quickly return home.

The results will have an interest in both the assessment on the management of post-stroke psychiatric disorders: distinguishing characteristics of depression and anxiety consecutive in this event in order to facilitate the diagnosis from the acute phase stroke and direct support. The symptomatological risk profiles can thus be detected and specific therapies on the prominent symptoms such disorders in the field of stroke may be proposed and / or developed.

Moreover, the results will enable a greener and more detailed understanding of the process connecting the individual coping strategies, post-stroke psychological problems and quality of life in various important time of the disease.

project interests Our project has several interests. First, it provides a longitudinal study tracking over the first months post-stroke, combining several complementary assessment methods that will enable a more comprehensive representation of psychological manifestations: standardized tools traditionally used and more environmentally friendly methods.

This design study should provide a better understanding of psychic and their development at key stages of life process for patients after stroke (hospitalization in another service, return home).

Several clinical implications are expected: develop prevention of post-stroke psychological problems by allowing the specific identification of depression and anxiety from the acute phase; identify targeted supported on the specifics of these disorders in the field of stroke; improve Supported favoring the development of coping strategies associated with long-term mental health and to reduce those associated with negative development; understand how these healthy patients after stroke and quickly return home, live these important steps to provide support tailored to suit their specific needs.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,
* first diagnosis of ischemic or hemorrhagic stroke,
* with a rapid recovery prognosis from hospitalization in intensive care (NIHSS score less than or equal to 6 at the output of the intensive care unit).

Exclusion Criteria:

* diagnosis of other somatic or neurological chronic,
* Current diagnosis of psychotic disorder or past,
* Diagnosis of dementia,
* Severe aphasia (NIHSS subscore),
* Visual or motor disabilities prevent participation in the study (subscores NIHSS),
* Reduced autonomy (Rankin score greater than 3).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Assessment the change of WHOQOL BREF (Life QUALITY) change | T1 (Day 0 outside the neurovascular unit).T2 (Month 2 after Cerebral Stoke). T3 (Month 4 After Cerebral Stoke)

SECONDARY OUTCOMES:
Assessment the change of MINI (Mini International Neuropsychiatric Inventory) score | T0 (Day 4-7 after Cerebral Stoke). T3 (Month 4 after Cerebral Stoke)
Assessment the change of MADRS (Montgoméry and Asberg Depression Rating Scale) score | T0 (Day 4-7 after Cerebral Stoke). T3 (Month 4 after Cerebral Stoke)
Assessment the change of HAM-A (Hamilton Anxiety Rating Scale) score | T0 (Day 4-7 after Cerebral Stoke). T3 (Month 4 after Cerebral Stoke)
Assessment the change of BDI-II (Beck Depression Inventory 2e ed) score | T1 (Day 0 outside the neurovascular unit).T2 (Month 2 after Cerebral Stoke). T3 (Month 4 After Cerebral Stoke)
Assessment the change of HADS (Hospital Anxiety Depression Scale) score | T1 (Day 0 outside the neurovascular unit).T2 (Month 2 after Cerebral Stoke). T3 (Month 4 After Cerebral Stoke)
Assessment the change of Brief-COPE score | T1 (Day 0 outside the neurovascular unit).T2 (Month 2 after Cerebral Stoke). T3 (Month 4 After Cerebral Stoke)
  This questionnaire assesses 14 separate dimensions of coping (two items per dimensions): active coping, planning, instrumental support, emotional support, expression of feelings, positive reinterpretation, acceptance, denial, blame, humor, religion, entertainment, substance use and disengagement Behavioural
Assessment the change of ESM score | T1 (Day 0 outside the neurovascular unit).T2 (Month 2 after Cerebral Stoke). T3 (Month 4 After Cerebral Stoke)
  These measures will be carried out via a smartphone app. Symptoms of depression and anxiety: the symptoms of depression and anxiety present in the DSM-IV-TR and show a variability in a day will be assessed dimensionally on a Likert scale 7 points. Eg for depression: sad mood, anhedonia, fatigue, difficulty concentrating, negative / pessimistic thoughts.
  Life events: questions will focus on the occurrence in the last three hours of events that have a positive impact on one hand, and negative on the other. Participants should indicate the specific areas of life for these events .
  strategies to adapt to stressful events: coping strategies will be evaluated by adapting the questions brief-COPE. Participants will indicate how they reacted to the negative event previously identified by selecting from a list of st

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu ZUBER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hopitalier Paris Saint Joseph Service de neurologie, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Alpers GW. Ambulatory assessment in panic disorder and specific phobia. Psychol Assess. 2009 Dec;21(4):476-85. doi: 10.1037/a0017489. PMID 19947782